CLINICAL TRIAL: NCT03481257
Title: Comparison of Shear Stress-induced Thrombotic and Thrombolytic Effect d Thrombolytic Effect Between Ticagrelor Versus Very Low Dose Rivaroxaban With Clopidogrel in Patients With Acute Coronary Syndrome
Brief Title: Comparison Between Ticagrelor Versus Very Low Dose Rivaroxaban With Clopidogrel
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, Principal Investigator, Seoul National University Hospital
Other Study IDs: 06-2017-086
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ticagrelor: ACS patients treated with aspirin (100mg/d) and ticagrelor (90mg bid)
- Clopidogrel + very low dose rivaroxaban: ACS patients treated with aspirin (100mg/d), clopidogrel(75mg/d) and very low dose rivaroxaban (2.5mg bid)

SUMMARY:
A total of 50 participants diagnosed with ACS (group A ticagrelor 180mg/d, n=25), group B (clopidogrel 75mg + rivaroxaban 5mg/ d, n=25)) were consecutively enrolled and treated with study drugs on top of aspirin (100mg/d) for 1 month. VerifyNow® and Global thrombosis test were performed at day 2 and 1 month after administration of study drugs. The investigators compared aspirin reaction unit (ARU) and P2Y12 reaction unit (PRU), occlusion time (OT) which reflects shear stress-induced thrombotic activity, and lysis time (LT) which showed endogenous lytic activity between the two strategies at both time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with acute coronary syndrome and underwent percutaneous coronary intervention

Exclusion Criteria:

* Patients administered with glycoprotein IIb/IIIa inhibitiors
* Patients with atrial fibrillation
* Patients with high risk of bleeding at the physician's discretion
* Patients with renal impairment (estimated GFR <30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-six patients from 452 patients who underwent percutaneous coronary intervention (PCI) due to ACS in Seoul National University Bundang Hospital. ( April 2017~ January 2018)
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-02-04 (Actual)

PRIMARY OUTCOMES:
Occlusion time | 1 month
  Global thrombosis test

SECONDARY OUTCOMES:
Lysis time | 1 month
  Global thrombosis test
Occlusion time | Day 2
  Global thrombosis test
Lysis time | Day 2
  Global thrombosis test
P2Y12 reaction unit | Day 2 and 1 month
  VerifyNow test
Aspirin reaction unit | Day 2 and 1 month
  VerifyNow test

OTHER OUTCOMES:
major adverse cardiovascular outcome | 1 month
  composites of cardiac death, myocardial infarction and target lesion revascularization
BARC bleeding | 1 month
  ARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided